CLINICAL TRIAL: NCT04160455
Title: Study of Autophagy and the Effects of GALIG Gene Products in HIV-1 Infected Patients Who Are Under Antiretroviral Therapy Since Primary-infection, Chronic Phase, or Never Treated.
Acronym: ATGALIG-HIV
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2019-03
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Autophagy; Galectins; HIV Infections; Highly Active Antiretroviral Therapy
Keywords: Antiretroviral therapy; basal autophagy; GALIG gene; HIV; apoptosis
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cohort A, group A1: 40 patients on suppressive antiretroviral therapy (HIV RNA <50 copies / ml for at least 4 years) initiated during the chronic phase : CD4 count less than 500 cells / ml at the time of inclusion in the study
  Interventions: Biological: expression of a panel
- Cohort A, group A2: 40 patients on suppressive antiretroviral therapy (HIV RNA <50 copies / ml for at least 4 years) initiated during the chronic phase: CD4 count above 500 cells / ml at the time of inclusion in the study
  Interventions: Biological: expression of a panel
- Cohort B: 20 patients on suppressive antiretroviral therapy (HIV RNA <50 copies / ml for at least 4 years) initiated since the primary-infection (within 4 months after acute infection)
  Interventions: Biological: expression of a panel
- Cohort C, group C1: 20 patients with detectable HIV RNA, naïve of antiretroviral, but who have an indication to start antiretroviral therapy: HIV diagnosis made during primary infection (within 4 months of infection)
  Interventions: Biological: expression of a panel
- Cohort C, group C2: 20 patients with detectable HIV RNA, naïve of antiretroviral, but who have an indication to start antiretroviral therapy: HIV diagnosis made during the chronic phase (more than 1 year after contamination), with CD4 count above 200 cells/ml at the time of inclusion in the study
  Interventions: Biological: expression of a panel
- Cohort C, group C3: 20 patients with detectable HIV RNA, naïve of antiretroviral, but who have an indication to start antiretroviral therapy: HIV diagnosis made during the chronic phase (more than 1 year after contamination), with CD4 count less than 200 cells/ml at the time of inclusion in the study
  Interventions: Biological: expression of a panel
- Cohort D: 20 patients who have undetectable plasma HIV RNA (HIV RNA <50 copies / ml ) without antiretroviral therapy, either spontaneously (HIV controllers or elite controllers) or after treatment interruption (post-treatment controllers).
  Interventions: Biological: expression of a panel

INTERVENTIONS:
Biological: expression of a panel — Quantify, by droplet digital PCR, the expression of a panel of 7 genes (+ GALIG) involved in autophagy2 on sub-populations (CD4+ and CD8+ lymphocytes and monocytes) after their sorting using magnetic bead cell then RNA extraction Evaluate, on a functional test (as previously described1), whether the observed expression dysregulation is associated with a deregulation of the autophagic function, whether constitutive or induced.

SUMMARY:
Little is known about autophagy during HIV infection. Recently, two different teams reported important dysfunctions of autophagy in HIV-infected patients despite sustained suppressive antiretroviral therapy. As altered autophagy is strongly linked to cellular senescence and chronic inflammation, two hallmarks of HIV-infected patients despite long-term suppressive antiretroviral therapy, it is important to improve our knowledge in the area.

Our main objective is to determine whether all or part of mononuclear cell subpopulations (CD4+ and CD8+ T lymphocytes, and monocytes) exhibit a defect in autophagy function in a cohort of HIV-infected patients who are virologically-controlled (plasma HIV RNA <50 copies / ml) either spontaneously (i.e. HIV controllers or post-treatment controllers) or after they started antiretroviral therapy at different time points (i.e. at the acute or chronic phases), as compared with a control group (i.e. uninfected healthy blood donors).

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Age >=18 years
* Man or woman
* Infected with HIV-1 (and not co-infected with HIV-2)
* Followed at Orleans' Regional Hospital
* Patient belonging to one of the predefined cohorts/groups (see below)
* Patient having provided a written consent

Specific profiles of HIV-infected patients for the ATGALIG-HIV study:

Cohort A: patients on suppressive antiretroviral therapy (HIV RNA <50 copies / ml for at least 4 years) initiated during the chronic phase, divided into 2 groups according to the following criteria:

* group A1: CD4 count less than 500 cells / ml at the time of inclusion in the study
* group A2: CD4 count above 500 cells / ml at the time of inclusion in the study Cohort B: patients on suppressive antiretroviral therapy (HIV RNA <50 copies / ml for at least 4 years) initiated since the primary-infection (within 4 months after acute infection)

Cohort C: patients with detectable HIV RNA, naïve of antiretroviral, but who have an indication to start antiretroviral therapy, divided into the following 3 groups:

* group C1: HIV diagnosis made during primary infection (within 4 months of infection)
* group C2: HIV diagnosis made during the chronic phase (more than 1 year after contamination), with CD4 count above 200 cells/ml at the time of inclusion in the study
* group C3: HIV diagnosis made during the chronic phase (more than 1 year after contamination), with CD4 count less than 200 cells/ml at the time of inclusion in the study Cohort D: patients who have undetectable plasma HIV RNA (HIV RNA <50 copies / ml ) without antiretroviral therapy, either spontaneously (HIV controllers or elite controllers) or after treatment interruption (post-treatment controllers)

Exclusion Criteria:

* Patient unable, according to the investigator, to meet the requirements of the protocol
* Pregnant or lactating woman
* Patient with a history of inflammatory bowel disease, malignancy, intestinal ischemia, malabsorption or other gastrointestinal dysfunction that, in the judgment of the investigator, could interfere with the interpretation of the results.
* Presence of coagulation abnormality or unexplained bleeding history
* Treatment with oral or injectable anticoagulant (curative or preventive)
* Patient covered by Article L.1121-5 to L.1121-8 and L.1122-1-2 of the French Public Health Code (including minors and protected adults)
* Patient under guardianship or curatorship
* Patient who uncovered by French health insurance Patient participating in another clinical trial, evaluating a treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV-1-infected adults (not co-infected with HIV-2), followed at the Infectious Diseases Department of Orleans' Regional Hospital and meeting the inclusion criteria, will be offered to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2029-11-07 (Estimated); Study Completion 2039-11-07 (Estimated)

PRIMARY OUTCOMES:
Quantify of a panel of genes involved in autophagy on sub-populations | Quantifications will be done once for all patients (Day 0), except in cohort C where they will be repeated after they started antiretroviral therapy (at month 1, 3, 6, 12 and 24)
  Quantify by droplet digital PCR, the expression of a panel of 7 genes (+ GALIG) involved in autophagy on sub-populations (CD4+ and CD8+ lymphocytes and monocytes) after their sorting using magnetic bead cell then RNA extraction
functional test on mononuclear cell subpopulations in the autophagy function | Quantifications will be done once for all patients (Day 0), except in cohort C where they will be repeated after they started antiretroviral therapy (at month 1, 3, 6, 12 and 24)
  Evaluate on a functional test whether the observed expression dysregulation is associated with a deregulation of the autophagic function, whether constitutive or induced.
Validation of the expression assays of genes involved in the autophagy function | Quantifications will be done once for all patients (Day 0), except in cohort C where they will be repeated after they started antiretroviral therapy (at month 1, 3, 6, 12 and 24)
  Validate the expression assays of genes involved in the autophagy process and the statistical analyzes obtained on PBMCs on a validation cohort.

SECONDARY OUTCOMES:
analyze regulatory markers on dysregulated gene promoters | Tests will be done once for all patients (Day 0), except in cohort C where they will be repeated after they started antiretroviral therapy (at month 1, 3, 6, 12 and 24)
  To analyze regulatory markers on dysregulated gene promoters, we will analyze and compare the epigenetic marks (acetylation and methylation of histones, DNA methylation) overall and on the promoter zones of autophagy genes which present an alteration of expression.
quantify the reservoir of virus and ongoing viral replication | Tests will be done once for all patients (Day 0), except in cohort C where they will be repeated after they started antiretroviral therapy (at month 1, 3, 6, 12 and 24)
  To quantify the reservoir of virus and ongoing viral replication, we will respectively evaluate the integrated viral DNA and the 2LTR circles levels.
analyze the phenotype of the PBMCs studied | Tests will be done once for all patients (Day 0), except in cohort C where they will be repeated after they started antiretroviral therapy (at month 1, 3, 6, 12 and 24)
  To analyze the phenotype of the PBMCs studied, whether HIV positive or negative, we will evaluate, by analysis of surface markers in flow cytometry:
  * Distribution of CD3+CD4+, CD3+CD8+, NK, B, NK-T and monocyte populations
  * Activation (HLA-DR and CD38 on T cells; HLA-DR, CD11b and CD16 on monocytes)
  * Senescence (CD57+ on CD8+ T cells, CD7- on CD4+ T cells)
  * Exhaustion (PD1 / CD279)
  * Distribution of memories, naive and effector CD4+ and CD8+ lymphocytes (CD45RA and CCR7 / CD197)
  * Proliferative capacity of PBMCs
Evaluation of the level of inflammation | Tests will be done once for all patients (Day 0), except in cohort C where they will be repeated after they started antiretroviral therapy (at month 1, 3, 6, 12 and 24)
  To assess the level of inflammation, we will dose the inflammatory cytokines present in the patients' serum and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent HOCQUELOUX, Dr, Principal Investigator — CHR d'orléans
Locations (1):
- CHU Orleans, Orléans, France

REFERENCES:
- [Background] Deeks SG, Lewin SR, Havlir DV. The end of AIDS: HIV infection as a chronic disease. Lancet. 2013 Nov 2;382(9903):1525-33. doi: 10.1016/S0140-6736(13)61809-7. Epub 2013 Oct 23. PMID 24152939
- [Background] Ipp H, Zemlin A. The paradox of the immune response in HIV infection: when inflammation becomes harmful. Clin Chim Acta. 2013 Feb 1;416:96-9. doi: 10.1016/j.cca.2012.11.025. Epub 2012 Dec 7. PMID 23228847
- [Background] Serrano A, El Haddad S, Moal F, Prazuck T, Legac E, Robin C, Brule F, Charpentier S, Normand T, Legrand A, Hocqueloux L, Mollet L. Dysregulation of apoptosis and autophagy gene expression in peripheral blood mononuclear cells of efficiently treated HIV-infected patients. AIDS. 2018 Jul 31;32(12):1579-1587. doi: 10.1097/QAD.0000000000001851. PMID 29734217
- [Result] Gomez-Mora E, Robert-Hebmann V, Garcia E, Massanella M, Clotet B, Cabrera C, Blanco J, Biard-Piechaczyk M. Brief Report: Impaired CD4 T-Cell Response to Autophagy in Treated HIV-1-Infected Individuals. J Acquir Immune Defic Syndr. 2017 Feb 1;74(2):201-205. doi: 10.1097/QAI.0000000000001201. PMID 27787338